CLINICAL TRIAL: NCT07404384
Title: Impact of Slow Breathing and Its Interaction With Psychological Variables From the Fear-Avoidance Model of Pain on Heart Rate Variability and Resistance Exercise Performance in Women With Fibromyalgia.
Brief Title: Slow Breathing and Resistance Exercise in Fibromyalgia
Acronym: Breath-fibro
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Asociación de Pacientes de Fibromialgia y Síndrome de Fatiga Crónica de Málaga (APAFIMA) (Unknown); Asociación de Fibromialgia y Síndrome de Fatiga Crónica de Málaga (AFIBROMA) (Unknown)
Responsible Party: Principal Investigator, Elena R. Serrano-Ibáñez, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UW-UMA_177-2025-H
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Fibromyalgia; Fibromyalgia Syndrome
Keywords: Slow Breathing; Diaphragmatic Breathing; Heart Rate Variability; Resistance Exercise; Fear-Avoidance Model; Central Sensitivity Syndrome; Exercise Performance; Pain Catastrophizing; Kinesiophobia
MeSH Terms: conditions — Fibromyalgia; Hypoventilation; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Three-arm parallel group design with 1:1:1 randomization to slow breathing with pacer, slow breathing without pacer, or spontaneous breathing control
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Slow Breathing with Visual Pacer (Experimental): Participants perform 8 minutes of paced slow breathing (6 breaths/min) with continuous visual guidance before resistance exercise test.
  Interventions: Behavioral: Slow Breathing with Visual Pacer
- Slow Breathing without Visual Pacer (Experimental): Participants perform 8 minutes of self-paced slow breathing (6 breaths/min target) after brief training, without continuous visual guidance, before resistance exercise test.
  Interventions: Behavioral: Slow Breathing without Visual Pacer
- Spontaneous Breathing (Experimental): Participants breathe naturally at their spontaneous rate for equivalent duration before resistance exercise test.
  Interventions: Behavioral: Spontaneous Breathing (Active Control)

INTERVENTIONS:
Behavioral: Slow Breathing with Visual Pacer — Participants receive brief training using a visual pacer displayed on computer screen showing a line that rises during inhalation and falls during exhalation. The pacing is set to 6 respiratory cycles per minute (4 seconds inhalation, 6 seconds exhalation). Participants place one hand below chest and abdomen to monitor diaphragmatic movement. After training, participants continue slow breathing with the visual pacer continuously displayed, maintaining the prescribed respiratory rate.
  Arms: Slow Breathing with Visual Pacer
Behavioral: Slow Breathing without Visual Pacer — Participants receive identical brief training using the visual pacer to learn the slow breathing pattern (6 cycles per minute: 4 seconds inhalation, 6 seconds exhalation). Hand placement below chest and abdomen to monitor diaphragmatic movement. After training, the visual pacer is removed and participants attempt to maintain the slow breathing pattern independently without external guidance.
  Arms: Slow Breathing without Visual Pacer
Behavioral: Spontaneous Breathing (Active Control) — Participants spend equivalent time breathing at their natural, spontaneous rate. They receive similar attention from evaluators but no specific breathing instructions. Participants are instructed to breathe normally at their usual pace and rhythm.
  Arms: Spontaneous Breathing

SUMMARY:
This randomized controlled trial investigates whether slow breathing techniques influence heart rate variability, exercise self-efficacy, and resistance exercise performance in women with fibromyalgia. Participants will be randomly assigned to one of three breathing conditions (slow breathing with visual pacer, slow breathing without pacer, or spontaneous breathing) before performing a biceps curl resistance exercise. The study will examine how breathing patterns interact with psychological variables (anxiety sensitivity, pain catastrophizing, pain hypervigilance, and kinesiophobia) to affect physiological and performance outcomes.

DETAILED DESCRIPTION:
Background: Fibromyalgia is considered one of the most representative central sensitivity syndromes, where central sensitization is the predominant characteristic. Resistance and strength training have demonstrated efficacy as therapeutic strategies for fibromyalgia patients. Slow breathing has been shown to reduce anxiety, perceived stress, and pain intensity while increasing heart rate variability (HRV), a biomarker of stress reactivity. The Fear-Avoidance Model of Pain demonstrates that anxiety sensitivity, pain catastrophizing, hypervigilance, and fear of pain/movement largely determine activity levels in chronic pain patients. However, no studies have examined how slow breathing interacts with these psychological variables to enhance resistance exercise performance in fibromyalgia patients.

Study Design: Single-session, three-arm randomized controlled trial with parallel group assignment.

Experimental Procedure:

Phase 1 - Baseline Assessment:

* Semi-structured interview for demographic and clinical information
* Administration of self-report questionnaires (detailed below)
* 5-minute baseline HRV measurement (seated, eyes open, spontaneous breathing)
* Respiration rate inferred from HRV

Phase 2 - Resistance Exercise Preparation:

* Determination of optimal weight for biceps curl exercise using submaximal protocol
* Warm-up: 3 minutes walking + 10 unloaded practice repetitions
* Progressive weight testing to determine 50% 1-RM equivalent

Phase 3 - Breathing Intervention (8 minutes): Participants randomly assigned to:

* Condition A: Slow breathing with visual pacer (6 breaths/min: 4-sec inhale, 6-sec exhale) displayed continuously
* Condition B: Slow breathing without pacer (same pattern, brief training then self-paced)
* Condition C: Spontaneous breathing at participant's natural rate
* HRV continuously recorded during all breathing conditions. Respiration rate inferred from HRV.

Phase 4 - Resistance Exercise Test:

* Biceps curl exercise at 50% estimated 1-RM
* Maximum repetitions to voluntary exhaustion
* Proper form maintained (back against wall, arms close to body, full range of motion)

Phase 5 - Post-Exercise Assessment:

* Immediate measurement of dependent variables (detailed below)
* 8 min. of rest
* HRV recording 5 min.

Safety Monitoring: Continuous observation by trained evaluators; clear stopping criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Female sex
2. Age ≥ 18 years
3. Medical diagnosis of fibromyalgia confirmed by physician
4. Capacity to understand and sign informed consent form
5. Fluency in spoken and written Spanish

Exclusion Criteria:

1. Current or past severe mental illness or neurodegenerative disease
2. Current treatment for oncological pathology, degenerative disease, or terminal illness
3. Musculoskeletal injury contraindicating biceps curl exercise
4. Connective tissue disease or arthritis
5. Inability to perform biceps curl exercise due to physical limitations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) - Change from Baseline | Measured: 5 min baseline, 8 min during breathing intervention, and 5 min post-exercise recovery.
  Root mean square of successive differences (RMSSD) in milliseconds
Number of Biceps Curl Repetitions | Immediately during the resistance exercise test (single session).
  Number of properly executed biceps curl repetitions at 50% estimated 1-RM performed to voluntary exhaustion with proper form maintained.

SECONDARY OUTCOMES:
Exercise-Related Self-Efficacy | Immediately post-exercise.
  Single-item 0-10 numeric rating scale.
Fatigue | Immediately post-exercise
  Borg Rating Of Perceived Exertion. Rating of perceived exertion is an outcome measure scale used to gauge one's exercise intensity without the need to rely on physiological parameters. The scale rates exertion from a scale of 6 (no exertion) to 20 (maximum effort).
Change in Current Pain Intensity | Immediately post-exercise
  Numeric Rating Scale (NRS) 0-10
Change in Anxiety | Immediately post-exercise.
  Numeric Rating Scale (NRS) 0-10
Perceived effort required to do the biceps exercise | Immediately post-exercise
  Numeric Rating Scale (NRS) 0-10.
Breathing Difficulty | Immediately after breathing intervention.
  Numeric Rating Scale (NRS) 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Czub, PhD, Principal Investigator — University of Wrocław; Rosa Esteve, PhD, Principal Investigator — University of Malaga; Elena R. Serrano-Ibáñez, PhD, Principal Investigator — University of Malaga; Joanna Piskorz, PhD, Principal Investigator — University of Wrocław
Locations (2):
- Spain (2):
  - Asociación de Fibromialgia y Síndrome de Fatiga Crónica de Málaga (AFIBROMA), Málaga, Málaga
  - Asociación de Pacientes de Fibromialgia y Síndrome de Fatiga Crónica de Málaga (APAFIMA), Málaga, Málaga

IPD SHARING:
Plan to Share IPD: Yes
We will share the joint database through a web link for public access.

REFERENCES:
- [Background] Yunus MB. Central sensitivity syndromes: a new paradigm and group nosology for fibromyalgia and overlapping conditions, and the related issue of disease versus illness. Semin Arthritis Rheum. 2008 Jun;37(6):339-52. doi: 10.1016/j.semarthrit.2007.09.003. Epub 2008 Jan 14. PMID 18191990
- [Background] Rogers AH, Farris SG. A meta-analysis of the associations of elements of the fear-avoidance model of chronic pain with negative affect, depression, anxiety, pain-related disability and pain intensity. Eur J Pain. 2022 Sep;26(8):1611-1635. doi: 10.1002/ejp.1994. Epub 2022 Jul 7. PMID 35727200
- [Background] Bamert M, Inauen J. Physiological stress reactivity and recovery: Some laboratory results transfer to daily life. Front Psychol. 2022 Aug 15;13:943065. doi: 10.3389/fpsyg.2022.943065. eCollection 2022. PMID 36046406
- [Background] da Silva JM, de Barros BS, Almeida GJ, O'Neil J, Imoto AM. Dosage of resistance exercises in fibromyalgia: evidence synthesis for a systematic literature review up-date and meta-analysis. Rheumatol Int. 2022 Mar;42(3):413-429. doi: 10.1007/s00296-021-05025-9. Epub 2021 Oct 15. PMID 34652480
- [Background] Goheen J, Anderson JAE, Zhang J, Northoff G. From Lung to Brain: Respiration Modulates Neural and Mental Activity. Neurosci Bull. 2023 Oct;39(10):1577-1590. doi: 10.1007/s12264-023-01070-5. Epub 2023 Jun 7. PMID 37285017
- [Background] Andrade A, de Azevedo Klumb Steffens R, Sieczkowska SM, Peyre Tartaruga LA, Torres Vilarino G. A systematic review of the effects of strength training in patients with fibromyalgia: clinical outcomes and design considerations. Adv Rheumatol. 2018 Oct 22;58(1):36. doi: 10.1186/s42358-018-0033-9. PMID 30657077